CLINICAL TRIAL: NCT00924586
Title: Study of ONO-1101 in Patients Scheduled for Multi-Slice Computed Tomography (CT), a Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Center Study
Brief Title: Study of ONO-1101 in Patients Scheduled for Multi-Slice Computed Tomography (CT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ONO-1101-27
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — landiolol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: ONO-1101
- E (Experimental)
  Interventions: Drug: ONO-1101

INTERVENTIONS:
Drug: ONO-1101 — Placebo for one minute IV
  Arms: P
Drug: ONO-1101 — 0.125 mg/kg for one minute IV
  Arms: E

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-1101 in patients scheduled for multi-slice CT, in a double-blind, randomized, placebo-controlled, parallel group, multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years old
* Heart rate ≥ 70beats/min and ≤ 90beats/min at entering the CT room and just before dosing organic nitrates.

Exclusion Criteria:

* Previous allergic reactions to contrast agent
* Renal failure
* Asthma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Image quality | one day

SECONDARY OUTCOMES:
Heart rate | 5 days maximum

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (2):
- Japan (2):
  - Kanto Region, Kanto
  - Kyushu Region, Kyushu